CLINICAL TRIAL: NCT03173794
Title: CommunityRx for Hunger: A Children's Hospital-Based Intervention to Support Caregivers in an African American Community
Brief Title: CommunityRx for Hunger: A Hospital-Based Intervention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This trial was a duplicate entry. Recruitment was never open and no participants were enrolled.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB17-0770
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Food Insecurity; Caregivers; Clinical Trial; Hunger; Health-Related Quality of Life; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Only (No Intervention): The control group will receive usual care, no CommunityRx-H intervention
- Usual Care and Intervention (Experimental): The intervention arm will receive the CommunityRx-H intervention, an information-based intervention that provides referrals to community resources
  Interventions: Other: CommunityRx-H

INTERVENTIONS:
Other: CommunityRx-H — CommunityRx-H has two components: (1) health-information technology (HIT) e-prescribing, and (2) a Community Resource Specialist (CRS). CommunityRx functions like an e-prescribing system: a HealtheRx "prescription" is automatically generated at the point of care. The HealtheRx provides referrals to food resources and federal nutrition assistance information tailored to the caregiver's address and proactive social support in the form of SMS-text message nudges from the CRS. Caregivers in the intervention arm are able to request information on resources not limited to food, including employment support, help paying rent or mortgage, etc. Nudges will promote caregiver self- and family management by increasing knowledge of and encouraging activation of community resources.
  Arms: Usual Care and Intervention

SUMMARY:
The goal of this research program is to reduce health disparities by deploying an information-based intervention to increase caregiver utilization of community-based food supports and satisfaction with care among food insecure caregivers of hospitalized children. We will conduct a randomized controlled trial to evaluate, versus usual care, the effects of the CommunityRx-H intervention on caregiver use of food resources (primary), caregiver patient satisfaction with care (primary), caregiver mental health-related quality of life (secondary), and caregiver household food security (secondary). The proposed research will yield an understanding of how to leverage a child's hospitalization to effectively intervene on the problem of food insecurity. Findings will inform the rapidly growing field of healthcare-based interventions to address health-related social needs.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* English-speaking
* Living in 1 of the 16 ZIP code target regions
* Self-identify as a primary caregiver of a child <18 years old hospitalized in CCH's general, intensive care or transplant units

Exclusion Criteria:

* Recollection of previous receipt of a HealtheRx

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in use of food resources | Baseline, 7 days, 30 days, 60 days, and 90 days
  Change in use of food resources will be measured using investigator-generated questions about use of the resources for self or others, sharing of information about the resources
Patient satisfaction with care | 7 days
  Patient satisfaction will be measured using the Patient Satisfaction Questionnaire (PSQ-18)

SECONDARY OUTCOMES:
Change from baseline in mental health-related quality of life | Baseline, 7 days, 30 days, 60 days, and 90 days
  Mental health-related quality of life will be measured using the Medical Outcomes Study Short Form-36
Change from baseline in household food insecurity | Baseline, 30 days, 60 days, and 90 days
  Household food insecurity will be measured using the 18-item Household Food Security Survey

OTHER OUTCOMES:
Change from baseline in caregiver stress | Baseline, 7 days, 30 days, 60 days, and 90 days
  Caregiver stress will be measured using the Perceived Stress Scale (PSS). Measure is included in the NIH Common Data Element Repository
Change from baseline in caregiver burden | Baseline, 7 days, 30 days, 60 days, and 90 days
  Caregiver burden will be measured using the Caregiver Burden Scale (CGBS). Measure is included in the NIH Common Data Element Repository
Change from baseline in caregiving self-efficacy | Baseline, 7 days, 30 days, 60 days, and 90 days
  Caregiver self-efficacy will be measured using General Self-Efficacy Scale (GSE). Measure is included in the NIH Common Data Element Repository
Change from baseline in contact Community Resource Navigator | Baseline, 7 days, 30 days, 60 days, and 90 days
  Change in contact with Community Resource Navigator will be measured using investigator-generated questions
Satisfaction with navigation | 7 days
  Patient satisfaction with logistical aspects of navigation will be measured using investigator-generated questions
Change in stigma during child's hospital stay | 7 days, 30 days, 60 days, 90 days
  Change in stigma will be measured using the Experiences of Discrimination Scale (EDS)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Lindau, MD, Principal Investigator — University of Chicago